CLINICAL TRIAL: NCT01259440
Title: Using Telemedicine to Improve Veteran Sleep Apnea Care
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PPO 10-101; H130392 (Other: VA San Diego Healthcare System)
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Sleep Apnea Syndromes
Keywords: Telemedicine; continuous positive airway pressure; treatment adherence
MeSH Terms: conditions — Sleep Apnea Syndromes; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Teleconferencing Care (Active Comparator): Video teleconferencing care
  Interventions: Behavioral: Video Teleconferencing Care
- Usual Care (Placebo Comparator): Usual Care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Video Teleconferencing Care — The core component of the VTC intervention is the frequent contact between patient and provider using a telemedicine system that allows for audio-visual communication.
  Arms: Video Teleconferencing Care
Behavioral: Usual Care — Consists of one week telephone call and one month clinic visit
  Arms: Usual Care

SUMMARY:
Obstructive sleep apnea (OSA) is highly prevalent in the Veteran population given the risk factors of male gender, being overweight, and increasing age. OSA is caused by upper airway obstruction, resulting in arousals from sleep and hypoxia. While continuous positive airway pressure (CPAP) is a highly efficacious treatment for OSA, compliance with treatment is suboptimal. Because research shows that adherence patterns are established early in treatment, we seek to use a technology that enables early and frequent productive interactions between patient and provider.

DETAILED DESCRIPTION:
Background:

Obstructive sleep apnea (OSA) is highly prevalent in the Veteran population given the risk factors of male gender, being overweight, and increasing age. OSA is caused by upper airway obstruction, resulting in arousals from sleep and hypoxia. While continuous positive airway pressure (CPAP) is a highly efficacious treatment for OSA, compliance with treatment is suboptimal. Because research shows that adherence patterns are established early in treatment, we seek to use a technology that enables early and frequent productive interactions between patient and provider

Objectives:

The objective of this proposal is to explore the feasibility and initially evaluate the potential efficacy of a video teleconferencing system for patients with Obstructive Sleep Apnea syndrome (OSA) that facilitates patient- centered, collaborative management for patients who are prescribed the gold-standard treatment, continuous positive airway pressure (CPAP).

Methods:

The evaluative aspect of this proposal was designed as a pilot randomized, controlled clinical trial of Video Teleconferencing (VTC) compared to Usual Care (UC). The key feature of the Video Teleconferencing intervention was the use of a telemedicine system that allows for audio/visual conferencing with the patient in their home environment from the start of treatment initialization. The provider is able provide more direct feedback to the patient based on the telemedicine interaction, and the patient benefits from increased contact with the provider. Specific inclusion and exclusion criteria included: age > 18 years; confirmed diagnosis of moderate-severe OSA; being newly prescribed CPAP therapy; having chronic symptoms as noted on screening symptom checklist; and fluency in English. Patients were recruited from the VA San Diego Healthcare System Pulmonary Sleep Clinic. Patients were enrolled for a 2-month time period. Groups were compared on quantitative and qualitative measures.

Status:

Study Complete

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Moderate to Severe Sleep Apnea
* Live in San Diego County
* Veteran

Exclusion Criteria:

* Previous use of positive pressure airway therapy
* Residence outside of San Diego county

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Stepnowsky, PhD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Video Teleconferencing Care | Usual Care
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video Teleconferencing Care | Usual Care | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (8.3) | 49.3 (11.3) | 52.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Treatment Adherence
Description: Nightly CPAP adherence measured over the two-month period .
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: hours/night
Arm/Group | Video Teleconferencing Care | Usual Care
Number analyzed (Participants) | 13 | 10
hours/night | 3.4 (2.4) | 3.6 (1.8)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Video Teleconferencing Care | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes